CLINICAL TRIAL: NCT05276999
Title: Rheumatic Heart Disease Community Streptococcal Treatment Program "RESET"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0026
Record Dates: First submitted 2022-01-14; First posted 2022-03-14 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Intervention Model Description: Pragmatic public health study to test an integrated strep education and treatment program to reduce echo-detected burden of RHD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Echocardiographic Screening of school age children (Experimental): Echocardiographic screening of school age children in Tororo and Iganga districts in Uganda to measure the prevalence of RHD before and two years after the deployment of an integrated strep infection education and treatment package.
  Interventions: Other: Healthcare provider education; Other: Community Awareness campaign
- Healthcare worker knowledge (Experimental): Health care worker representatives from 101 facilities (n=101) will participate in primary educational workshops in identifying and treating GAS pharyngitis.
  Interventions: Other: Healthcare provider education
- Health seeking behavior in the community (Experimental): To increase health seeking behavior for sore throat thorough a multifaceted community awareness campaign that includes school based education, VHT lead education, education of patients seeking evaluation of sore throat at HC, and public service announcements
  Interventions: Other: Community Awareness campaign

INTERVENTIONS:
Other: Healthcare provider education — Mix of training and educational activities within the district continuing medical education system targeting community health workers and frontline providers focused on the importance of sore throat and it's link to RHD, clinical guidelines to differentiate patients at high or low risk for GAS pharyngitis and guideline based care for treating GAS pharyngitis
  Arms: Echocardiographic Screening of school age children; Healthcare worker knowledge
Other: Community Awareness campaign — A district wide public health campaign to increase community awareness of sore throat, including school based education, VHT community sensitization, education of parents and patients, radio messaging, posters, signs and billboards.
  Arms: Echocardiographic Screening of school age children; Health seeking behavior in the community

SUMMARY:
The primary objective of this study is to determine the impact of a pragmatic RHD primary prevention program in Uganda.

The secondary Objective are as follow:

1. To improve guideline-based care for sore throat through frontline healthcare provider education on clinical decision rules and guideline-based primary prevention.
2. To increase health seeking behavior for sore throat thorough a multifaceted community awareness campaign.

DETAILED DESCRIPTION:
Our intervention is designed as a service-oriented plan to be implemented through the primary healthcare structure and facilities of both the national health and private system. Additional support will come from the education system, with participation from schools, teachers, patients, patient families, and the public. Our intervention will focus on two of the more easily rectified impediments to primary prevention, namely (1) poor uptake of guideline-based treatments for Group A Streptococcal (GAS) pharyngitis and (2) low levels of public awareness of the importance of sore throat care and treatment.

ELIGIBILITY:
Inclusion Criteria:

• Has agreed to participate in the study via the study's informed consent/assent process.

Exclusion Criteria:

* Known history of ARF or RHD
* Any known co-morbid conditions (HIV, renal deficiencies, severe malnutrition,
* among others) that have resulted in prescription of regular antibiotic prophylaxis
* Structural or functional cardiac defects, other than those consistent with RHD, that were known prior to or detected through echo screening (except patent foramen ovale, small atrial septal defect, small ventricular septal defect, small patent ductus arteriosus).

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66123 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Determination of Echocardiography prevalence of RHD among children 5-15 years old | 2 year endpoint
  Echocardiography screening of school age children in Uganda to determine prevalence of RHD prior to and 2 years post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z Beaton, Principal Investigator — Cincinnati Chidren's hospital
Locations (1):
- Uganda Heart Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No